CLINICAL TRIAL: NCT01993043
Title: Comparison of Vision and Development Outcomes in Laser- and Bevacizumab-Treated Infants With Retinopathy of Prematurity
Brief Title: 39946-I Laser and Bevacizumab Treatment for Retinopathy of Prematurity
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Lingkun Kong, Principal Investigator, Baylor College of Medicine
Other Study IDs: H-29628
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: ROP Threshold
Keywords: ROP; Bevacizumab; Laser; Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
Retinopathy of prematurity (ROP) is a leading cause of childhood blindness. Vascular endothelium growth factor (VEGF) is an important component of this disease. The goal of treatment is to reduce the production of VEGF in the immature retina and to eliminate the abnormal growth of new vessels. Currently, laser photocoagulation of the peripheral avascular retina is the treatment standard. Intravitreal injection of anti-VEGF antibody Bevacizumab (IVB) has been used clinically off-label as an alternative therapy. However, VEGF is important for the development of neurons and vessels in the systemic organs in premature infants. Pharmaceutical study showed that IVB was absorbed into the bloodstream. It is unclear if the systemic absorption of Bevacizumab is dose related, and the short and longterm effects on ocular and systemic systems, especially neurological development. In this study, our goals are to establish the pharmacokinetics of Bevacizumab in the premature infant and to compare the short and long-term vision and neurodevelopmental outcomes of infants treated with IVB compared to laser ROP.

DETAILED DESCRIPTION:
This study will enroll preterm infants who were scheduled to receive treatment for ROP by laser or Bevacizumab. We will observe the patients in the hospital for the cure of ROP until 54 weeks' postmenstrual age. We will check the changes of chemicals in the blood and observe short-term and long-term effects on visual system, brain and other body organs. Descriptive statistics from a two sample t-test or Fisher's exact test will be used to compare the short and long-term vision and neurological development outcomes. We predefined a statistical significance level p=0.05.

ELIGIBILITY:
Inclusion Criteria:

Premature infants who were scheduled to receive laser or BEvacizumab treatment for type I ROP .

Exclusion Criteria:

1. Have unilateral or Bilateral ROP Stage 4 or 5 ROP;
2. Lack of signed consent by the parent or legal guardian.

Ages: 30 Weeks to 40 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Premature infants
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-10; Primary Completion 2020-10 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Vision | 5 years
  Visual acuity will be measured at age of 3 and 5 years with HOTV card.

SECONDARY OUTCOMES:
The changes of neurodevelopment outcome from birth to 5 years of age | 1 to 5 years old
  Neurodevelopmental assessments will be performed by board-certified, developmental-behavioral pediatric and neurodevelopmental disability pediatricians. Each neurodevelopmental assessment includes a developmental history, direct behavioral observations, and direct developmental testing using the Revised Gesell Developmental Schedules; the Motor Quotient will be used to assess gross motor development; and the Capute Scales will be used used to assess non-verbal, visual-motor problem-solving development and speech and language development.

CONTACTS AND LOCATIONS:
Overall Officials: Lingkun Kong, MD, Ph.D, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Baylor College of Medicine, Houston, Texas
  - TTUHSC, Lubbock, Texas